CLINICAL TRIAL: NCT00885105
Title: Evaluation of Serologic Responses to Fluzone® in Infants ≥ 6 Months of Age Who Did or Did Not Receive Fluzone® Vaccine at 2 Months of Age
Brief Title: Evaluation of Responses to Fluzone® in Infants ≥ 6 Months of Age Who Did or Did Not Receive Fluzone® at 2 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC32
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Results first posted 2010-01-01 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Fluzone® vaccine; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluzone® Vaccine-Primed Group (Experimental): Participants received 2 doses of Fluzone® vaccine at 2 months (in Study GRC 27)
  Interventions: Biological: Influenza Virus Vaccine
- Influenza Vaccine-Naive Group (Active Comparator): Participants who have never received influenza vaccine (and not in Study GRC27)
  Interventions: Biological: Influenza Virus Vaccine

INTERVENTIONS:
Biological: Influenza Virus Vaccine — 0.25 mL, Intramuscular
  Other Names: Fluzone® 2005-2006 Pediatric Formulation
  Arms: Fluzone® Vaccine-Primed Group
Biological: Influenza Virus Vaccine — 0.25 mL, Intramuscular
  Other Names: Fluzone® 2005-2006 Pediatric Formulation
  Arms: Influenza Vaccine-Naive Group

SUMMARY:
The study is to compare the 2 Groups with respect to antibody responses to inactivated influenza vaccine.

Observational Objectives:

* To describe the percentage of participants with protective Hemagglutinin (HAI) antibody titers to each of the 3 vaccine antigens in both study groups following each vaccination.
* To describe the HAI geometric mean titer (GMTs) to each of the 3 vaccine antigens in both study groups following each vaccination.
* To describe the safety of the 2005-2006 pediatric formulation of Fluzone® vaccine in both study groups.

DETAILED DESCRIPTION:
This is a descriptive study that will provide preliminary comparative information about the safety and immunogenicity of Fluzone® vaccine among children who were given Fluzone® vaccine at 2 months of age (Study GRC27 NCT00858468)and those who never received influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Participant is between 6 and 10 months of age on the day of inclusion (has reached 6-month but has not reached 11-month anniversary of birth).
* Available for the duration of the study.
* Born at full term of pregnancy (≥ 36 weeks) with a birth weight ≥ 2.5 kg
* Parent/legal acceptable representative willing and able to provide informed consent.
* Parent/legal acceptable representative able to attend all scheduled visits and comply with all trial procedures.
* Parent/legal acceptable representative willing to permit venipuncture for purposes of collecting a blood sample.
* Previously enrolled in the 2-month-old group in Study GRC27 or approved by sponsor for enrollment as control.

Exclusion Criteria:

* Reported allergy to egg proteins, chicken proteins, or any other constituent of Fluzone vacccine.
* Previous history of influenza vaccination (Group 2 subjects only).
* Receipt of any vaccine in the 14 days prior to enrollment.
* An acute illness with or without fever (rectal temperature ≥ 38.0 °C [or ≥100.4 °F]) in the 72 hours preceding enrollment in the trial.
* Known bleeding disorder.
* Participation in any other interventional (e.g., vaccine, drug) clinical trial (except Study GRC27) within 30 days prior to enrollment, or planned participation in another interventional clinical trial prior to termination of the subject's participation in this study.
* Known or suspected impairment of immunologic function or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay, neurologic disorder, or seizure disorder.
* Chronic medical, congenital or developmental disorder that could interfere with trial conduct or completion.
* Known human immunodeficiency virus (HIV)-positive or hepatitis B surface antigen (HBsAg)-positive mother.
* Known HIV, hepatitis B, or hepatitis C infection.
* Receipt of blood or blood-derived products within the past 2 months.
* Prior history of Guillain-Barré syndrome.
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 242 (Actual)
Dates: Start 2005-10; Primary Completion 2006-01 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (6):
- United States (6):
  - Little Rock, Arkansas
  - Marietta, Georgia
  - Durham, North Carolina
  - Dayton, Ohio
  - Pittsburgh, Pennsylvania
  - Seattle, Washington

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 17 October 2005 to 05 January 2006 at 7 medical centers in the US.
Pre-assignment Details: A total of 242 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Fluzone® Vaccine-Primed Group: Participants had received 2 doses of Fluzone® vaccine at age 2 to 3 months; they received 2 doses of Fluzone® 2005-2006 pediatric formulation at age 6 to 11 months.
- Influenza Vaccine-Naive Group: Participants had never previously received influenza vaccine, they received 2 doses of Fluzone® 2005-2006 pediatric formulation at age 6 to 11 months.
Period: Overall Study
Arm/Group | Fluzone® Vaccine-Primed Group | Influenza Vaccine-Naive Group
Started | 112 | 130
Completed | 111 | 120
Not Completed | 1 | 10
Not completed — Withdrawal by Subject | 0 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone® Vaccine-Primed Group | Influenza Vaccine-Naive Group | Total
Number analyzed (Participants) | 112 | 130 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 112 | 130 | 242
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 7.29 (1.1) | 7.28 (1.47) | 7.28 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 60 | 113
  Male | 59 | 70 | 129
Region of Enrollment [Number; unit: participants]
  United States | 112 | 130 | 242

OUTCOME MEASURES:

1. Primary Outcome: Summary of Influenza Seroprotection Post-vaccination With Fluzone® Vaccine.
Description: Seroprotection was defined as a Reciprocal Hemagglutination Inhibition Titers of ≥ 40 Post-vaccination with Fluzone® Vaccine.
Time Frame: Day 28 Post-vaccination
Population: Hemagglutination inhibition titers to the Influenza vaccine antigens were assessed in the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone® Vaccine-Primed Group | Influenza Vaccine-Naive Group
Number analyzed (Participants) | 51 | 51
Percentage of Participants
  A/New Caledonia/20/99 Post-Dose 1 | 44 | 34
  A/New York/55/2004 Post-Dose 1 | 31 | 74
  B/Jiangsu/310/2003 Post-Dose 1 | 22 | 6
  A/New Caledonia/20/99 Post-Dose 2 | 69 | 86
  A/New York/55/2004 Post-Dose 2 | 84 | 100
  B/Jiangsu/310/2003 Post-Dose 2 | 28 | 47

2. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition Antibody Titers Post-Vaccination With Fluzone® Vaccine.
Description: Antibodies against Influenza virus in Fluzone® Vaccine determined by the Hemagglutination inhibition (HAI) assay method.
Time Frame: Day 28 Post-vaccination
Population: Geometric Mean Titers to the Influenza vaccine antigens were assessed in the per-protocol immunogenicity population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone® Vaccine-Primed Group | Influenza Vaccine-Naive Group
Number analyzed (Participants) | 51 | 51
Titers
  A/New Caledonia/20/99 Post-Dose 1 | 30.5 [22.3 to 41.8] | 18.9 [14.1 to 25.4]
  A/New York/55/2004 Post-Dose 1 | 21.4 [15.7 to 29.3] | 65.6 [47.7 to 90.2]
  B/Jiangsu/310/2003 Post-Dose 1 | 13.2 [9.89 to 17.6] | 6.2 [5.27 to 7.29]
  A/New Caledonia/20/99 Post-Dose 2 | 38.1 [29.6 to 49.2] | 104 [77.1 to 139]
  A/New York/55/2004 Post-Dose 2 | 78.9 [61.3 to 102] | 277 [223 to 346]
  B/Jiangsu/310/2003 Post-Dose 2 | 20.7 [16.1 to 26.6] | 23.9 [18.2 to 31.3]

3. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Pertussis, Tetanus, Diphtheria, and Haemophilus Influenzae, Antigens Post-vaccination With Fluzone® Vaccine.
Description: Antibodies against Pertussis, Tetanus, and Haemophilus influenzae antigens were determined by an indirect Enzyme linked immunosorbent assay (ELISA).
  Anti-diphtheria antibody response was measured by the Vero Cells - diphtheria toxin challenge method.
  The serological determinations of total anti-PRP antibody was performed using a Farr-type radioimmunoassay.
Time Frame: Day 28 Post-vaccination
Population: GMTs to the Pertussis, Tetanus, Diphtheria and Haemophilus Influenzae antigens were assessed in the per-protocol immunogenicity population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone® Vaccine-Primed Group | Influenza Vaccine-Naive Group
Number analyzed (Participants) | 94 | 104
Titers
  Pertussis Toxoid (EU/mL) | 57.9 [47.9 to 69.9] | 69.5 [57.6 to 83.7]
  Filamentous Hemagglutinin (EU/mL) | 37.3 [29.5 to 47.1] | 47.3 [37.9 to 59.0]
  Pertactin (EU/mL) | 22.0 [16.8 to 28.8] | 33.6 [26.1 to 43.2]
  Fimbriae Types 2 and 3 (EU/mL) | 26.7 [18.1 to 39.5] | 11.6 [7.76 to 17.4]
  Diphtheria (IU/mL) | 0.230 [0.180 to 0.294] | 0.251 [0.191 to 0.329]
  Tetanus (IU/mL) | 0.976 [0.694 to 1.37] | 0.980 [0.720 to 1.33]

4. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Polyribosylribitol Phosphate and Pneumococcal Antibodies After Concomitant Vaccination With Fluzone® Vaccine.
Description: Human antibodies to Streptococcus pneumoniae (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) were determined by an Enzyme linked immunosorbent assay (ELISA).
Time Frame: Day 28 post-vaccination
Population: Geometric Mean Titers (GMTs) for Polyribosylribitol Phosphate and Pneumococcal antibodies were determined in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone® Vaccine-Primed Group | Influenza Vaccine-Naive Group
Number analyzed (Participants) | 91 | 97
Titers
  Polyribosylribitol Phosphate (mcg/mL) | 1.69 [1.16 to 2.46] | 2.12 [1.49 to 3.02]
  Pneumococcal 4 (mcg/mL) | 1.02 [0.854 to 1.22] | 0.956 [0.781 to 1.17]
  Pneumococcal 6B (mcg/mL) | 1.14 [0.906 to 1.44] | 1.24 [0.949 to 1.61]
  Pneumococcal 9V (mcg/mL) | 0.974 [0.812 to 1.17] | 1.20 [0.981 to 1.46]
  Pneumococcal 14 (mcg/mL) | 4.98 [4.12 to 6.03] | 5.54 [4.56 to 6.74]
  Pneumococcal 18C (mcg/mL) | 0.783 [0.646 to 0.950] | 0.790 [0.644 to 0.970]
  Pneumococcal 19F (mcg/mL) | 1.49 [1.27 to 1.74] | 1.26 [1.05 to 1.51]
  Pneumococcal 23F (mcg/mL) | 0.920 [0.737 to 1.15] | 1.00 [0.779 to 1.29]

5. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Polio Antibodies After Concomitant Vaccination With Fluzone® Vaccine.
Description: Antibodies to polio viruses were measured by a serum neutralization assay.
Time Frame: Day 28 post-vaccination
Population: Geometric Mean Titers (GMTs) for the Polio antibodies were determined in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone® Vaccine-Primed Group | Influenza Vaccine-Naive Group
Number analyzed (Participants) | 94 | 104
Titers
  Polio Type 1 (1/dil) | 555 [415 to 742] | 1072 [814 to 1411]
  Polio Type 2 (1/dil) | 356 [268 to 474] | 550 [411 to 736]
  Polio Type 3 (1/dil) | 394 [282 to 551] | 571 [397 to 822]

6. Other Pre Specified Outcome: Percentage of Participants With Solicited Injection Site and Systemic Reactions Post-vaccination With Fluzone® Vaccine.
Description: Solicited injection site reactions: Tenderness, erythema and swelling. Solicited systemic reactions: Fever (temperature), vomiting, abnormal crying, drowsiness, loss of appetite, and irritability.
Time Frame: Days 0 up to 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone® Vaccine-Primed Group | Influenza Vaccine-Naive Group
Number analyzed (Participants) | 112 | 130
Percentage of Participants
  Any Solicited Injection Site Reaction Post-Dose 1 | 45 | 42
  Any Tenderness | 40 | 40
  Grd 3 Tenderness (injected limb movement reduced) | 1 | 1
  Any Redness (> 0.5 cm) | 11 | 14
  Grade 3 Redness (≥ 5.0 cm) | 2 | 1
  Any Swelling (> 0.5 cm) | 9 | 7
  Grade 3 Swelling (≥ 5.0 cm) | 1 | 0
  Any Solicited Injection Site Reaction Post-Dose 2 | 36 | 34
  Any Tenderness | 34 | 28
  Grd 3 Tenderness (injected limb movement reduced) | 1 | 0
  Any Redness (> 0.5 cm) | 12 | 10
  Grade 3 Redness ≥ 5.0 cm) | 0 | 0
  Any Swelling (> 0.5 cm) | 10 | 5
  Grade 3 Swelling (≥ 5.0 cm) | 1 | 0
  Any Solicited Injection Site Reaction - Any Dose | 51 | 51
  Any Tenderness | 48 | 45
  Grd 3 Tenderness (injected limb movement reduced) | 2 | 1
  Any Redness (> 0.5 cm) | 16 | 19
  Grade 3 Redness (≥ 5.0 cm) | 2 | 1
  Any Swelling (> 0.5 cm) | 13 | 10
  Grade 3 Swelling (≥ 5.0 cm) | 1 | 0
  Any Solicited Systemic Reaction Post-Dose 1 | 79 | 82
  Any Fever | 25 | 25
  Grade 3 Fever ≥ 103.3 ºF) | 0 | 1
  Any Vomiting | 14 | 7
  Grade 3 Vomiting (≥ 6 episodes per 24 hours) | 1 | 0
  Any Abnormal Crying | 46 | 32
  Grade 3 Abnormal Crying (> 3 hours) | 5 | 1
  Any Drowsiness | 47 | 45
  Grade 3 Drowsiness (difficulty waking up) | 1 | 1
  Any Loss of Appetite | 39 | 33
  Grd 3 Loss of Appetite (refuses ≥ 3 or most feeds) | 1 | 0
  Any Irritability | 65 | 63
  Grade 3 Irritability (inconsolable) | 2 | 1
  Any Solicited Systemic Reaction Post-Dose 2 | 64 | 62
  Any Fever | 14 | 14
  Grade 3 Fever (≥ 103.3 ºF) | 1 | 2
  Any Vomiting | 8 | 12
  Grade 3 Vomiting (≥ 6 episodes per 24 hours) | 0 | 3
  Any Abnormal Crying | 39 | 26
  Grade 3 Abnormal Crying (> 3 hours) | 2 | 3
  Any Drowsiness | 29 | 34
  Grade 3 Drowsiness (difficulty waking up) | 0 | 1
  Any Loss of Appetite | 29 | 28
  Grd 3 Loss of Appetite (refuses ≥ 3 or most feeds) | 0 | 1
  Any Irritability | 56 | 43
  Grade 3 Irritability (inconsolable) | 3 | 3
  Any Solicited Systemic Reaction - Any Dose | 86 | 90
  Any Fever | 32 | 34
  Grade 3 Fever (≥ 103.3 ºF) | 1 | 2
  Any Vomiting | 20 | 16
  Grade 3 Vomiting (≥ 6 episodes per 24 hours) | 1 | 2
  Any Abnormal Crying | 55 | 45
  Grade 3 Abnormal Crying (> 3 hours) | 6 | 3
  Any Drowsiness | 53 | 53
  Grade 3 Drowsiness (difficulty waking up) | 1 | 2
  Any Loss of Appetite | 52 | 43
  Grd 3 Loss of Appetite (refuses ≥ 3 or most feeds) | 1 | 1
  Any Irritability | 76 | 71
  Grade 3 Irritability (inconsolable) | 4 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 8 months. Six months post-vaccination 2
Arm/Group | Fluzone® Vaccine-Primed Group | Influenza Vaccine-Naive Group
Serious Adverse Events (participants affected / at risk) | 5/112 | 1/130
Other Adverse Events (participants affected / at risk) | 57/112 | 56/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone® Vaccine-Primed Group (N=112) | Influenza Vaccine-Naive Group (N=130)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 (0) | 1 (3)
Deafness bilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone® Vaccine-Primed Group (N=112) | Influenza Vaccine-Naive Group (N=130)
Conjunctivitis (Eye disorders) | 5 (5) | 7 (9)
Pyrexia (General disorders) | 8 (8) | 6 (6)
Bronchiolitis (Infections and infestations) | 5 (5) | 8 (8)
Croup infectious (Infections and infestations) | 7 (7) | 2 (2)
Otitis media (Infections and infestations) | 30 (34) | 30 (31)
Upper respiratory tract infection (Infections and infestations) | 20 (21) | 24 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 12 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications